CLINICAL TRIAL: NCT04582864
Title: A Phase 2 Trial Evaluating the Efficacy of Flotetuzumab (MGD006) for Relapsed Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) Following Allogeneic Hematopoietic Cell Transplantation (Allo-HCT)
Brief Title: Flotetuzumab for Relapsed Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) Following Allogeneic Hematopoietic Cell Transplantation (Allo-HCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor is no longer supporting the drug
Sponsor: Washington University School of Medicine (Other)
Collaborators: MacroGenics (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202011122; 5P50CA171963 (NIH)
Record Dates: First submitted 2020-09-25; First posted 2020-10-12 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Relapsed Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Flotetuzumab (Experimental): * Will start on cycle 1 day 1 on the dose escalation ramp schedule of flotetuzumab as a continuous intravenous (IV) infusion. Patients will be initiated at 30 ng/kg/day and have their dose increased daily to a target goal of 500 ng/kg/day by day 7
  * Patients will continue on flotetuzumab at 500 ng/kg/day for the remaining 21 days of the 28 day cycle.
  * On cycle 1 day 28, patients will undergo bone marrow biopsy for assessment of disease status. Patients who have achieved a CR/CRi will proceed to a second cycle per protocol, while patients with a PR or SD or better may proceed to cycle 2 with permission of the investigator. Patients with available donor lymphocytes may receive DLI concurrently with flotetuzumab during Cycle 1 and/or Cycle 2.
  Interventions: Drug: Flotetuzumab; Procedure: Donor lymphocyte infusion

INTERVENTIONS:
Drug: Flotetuzumab — Will be provided by MacroGenics Inc.
  Other Names: MGD006
Procedure: Donor lymphocyte infusion — DLI represents a non-specific form of adoptive cell therapy which involves infusion of a pool of allogeneic immune cells, including CD4+ T cells, CD8+ T cells, regulatory T cells (T Regs), natural killer (NK) cells and professional antigen presenting cells.
  Other Names: DLI

SUMMARY:
The investigators hypothesize that flotetuzumab for relapsed AML following allo-HCT will be safe, tolerable and may facilitate preferential immune effector cell retargeting of leukemic cells resulting in improved patient outcomes. Furthermore, administration of a donor lymphocyte infusion (DLI) (if available) in combination with flotetuzumab will be safe, tolerable and may provide additional therapeutic efficacy.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Histologically or cytologically confirmed relapsed acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS), including any AML subtype, except acute promyelocytic leukemia (APL), and including AML that has evolved from a previous MDS or MPN.
* Patients must have peripheral blast count ≤ 20,000/mm3. Use of hydroxyurea to control blast count is permitted.
* Patients must be status post allo-HCT (including: matched related, matched unrelated, haploidentical, mismatched unrelated; and cord blood HCT).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* Adequate organ function, defined as:

  * Hepatic transaminase (both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤2.5 times the institutional upper limit of normal (ULN),
  * Total bilirubin level ≤1.5 times the ULN (unless the patient has a history of Gilbert's Syndrome, in which case, total bilirubin must be ≤2.5 times the ULN),
  * Creatinine clearance of ≥50 ml/min
  * Adequate organ reserve including cardiovascular (ejection fraction within institutional normal limits), pulmonary (baseline pulmonary function test [PFT]: carbon monoxide diffusion capacity in the lung [DLCO] > 50%, forced expiratory volume in 1 second [FEV1] > 70%), renal, and hepatic functioning sufficient, in the judgment of the Investigator, to undergo therapy.
  * Normal thyroid function or stable thyroid tests on supplementation, except euthyroid sick syndrome.
* Recovery from toxicities of clinical consequence attributed to previous chemotherapy to CTCAE v4.0 Grade ≤ 1 (i.e., certain toxicities such as alopecia will not be considered in this category).
* Female patients of childbearing potential must test negative for pregnancy at enrollment and during the study. Sexually active women of child-bearing potential, unless surgically sterile, must be willing to use a highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1% per year) such as implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs) or vasectomized partner. Male patients with partners of childbearing potential must be either vasectomized or agree to use a condom in addition to having their partners use another method of contraception resulting in a highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1% per year) such as implants, injectables, combined oral contraceptives, or IUDs. Patients should not have sexual intercourse with females who are either pregnant or lactating without a condom. Contraception should be employed from the time of consent through 12 weeks after MGD006 administration. Patients should also abstain from sperm/egg donation during the course of the study.
* Able to have corticosteroids weaned to ≤0.5mg/kg prednisone/day (or equivalent)
* Able to have non-steroidal immunosuppression discontinued, including:

  * mycophenolate (MMF)
  * calcineurin inhibitors (tacrolimus, cyclosporine)

    **calcineurin inhibitors must be able to be discontinued at least 14 days prior to enrolling on study.
  * JAK inhibitors (ruxolitinib)
  * MTOR inhibitors (sirolimus)
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document

Recipient Exclusion Criteria:

* Active GVHD requiring systemic immunosuppression with more than 0.5 mg/day prednisone
* Currently receiving any other investigational agents.
* Any active untreated autoimmune disorders (with the exception of vitiligo, resolved childhood atopic dermatitis, prior Grave's disease now euthyroid clinically and with stable supplementation).
* Second primary malignancy that requires active therapy (adjuvant hormonal therapy is allowed).
* Antitumor therapy (chemotherapy, radiotherapy, antibody therapy, molecular- targeted therapy, retinoid therapy, or investigational agent) within 5 half-lives of Cycle 1 Day 1
* At the time of study entry, steroids >0.5mg/kg of prednisone or equivalent (except steroid inhaler, nasal spray or ophthalmic solution which are allowed).
* Use of immunosuppressant medications (other than steroids as noted) in the 2 weeks prior to study drug administration (Cycle 1 Day 1).
* Isolated extramedullary relapse (i.e., no evidence of bone marrow involvement).
* Known central nervous system (CNS) leukemia. Patients with suspected CNS leukemia must be evaluated by lumbar puncture and be free of CNS disease prior to study entry. Previously treated CNS leukemia is allowed provided adequate treatment has been provided and the patient is free of CNS disease.
* Any medical or psychiatric condition limiting full compliance or increasing the safety risk, at the discretion of the PI, such as:

  * active uncontrolled infection (including, but not limited to viral, bacterial, fungal, or mycobacterial infection),
  * known human immunodeficiency virus infection,
  * known, active, or chronic hepatitis B or C infection (appropriately treated HBV/HCV infections with documented clearance of viral titer are allowed),
  * Grade 3 or 4 bleeding,
  * significant pulmonary compromise including chronic supplemental oxygen use, history of non-infectious pneumonitis (including radiation pneumonitis), pulmonary fibrosis, or severe chronic obstructive pulmonary disease (COPD),
  * uncontrolled (persistent) hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 100 mm Hg
  * clinically significant arrhythmia, clinically significant baseline QTcF >480 msec,
  * unstable angina,
  * recent myocardial infarction within 6 months prior to study drug administration (Cycle 1 Day 1),
  * clinically significant heart disease, such as, congestive heart failure, history of pericarditis, myocarditis,
  * history of stroke or transient ischemic event within 3 months prior to study drug administration (Cycle 1 Day 1),
  * untreated pulmonary embolism, or non-catheter-related deep-vein thrombosis in the 3 months prior to study drug administration (Cycle 1 Day 1),
  * pregnancy, or breast feeding,
  * major surgery or trauma within 4 weeks before enrollment.
* Known hypersensitivity to murine, yeast, or recombinant proteins; polysorbate 80; recombinant human serum albumin; benzyl alcohol; or any excipient contained in the MGD006 drug formulation.
* Dementia or altered mental status that would preclude sufficient understanding to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Christopher, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared with other researchers.
Time Frame: From 2 years to 10 years after accrual closure
Access Criteria: IPD will be shared in de-identified form with investigators whose proposed use of the data has been approved by an independent review committee for that purpose.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flotetuzumab
Started | 11
Completed | 8
Not Completed | 3
Not completed — Did not complete cycle 1 due to disease progression | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 65 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Measured by Number of Participants With CR(Mrd), CR, and CRi
Description: * Complete remission without minimal residual disease (CRmrd): CR with negativity for a genetic marker by RT-qPCR, or CR with negativity by MFC
  * Complete remission (CR): Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0 × 10^9/L (1000/µL); platelet count ≥100 × 10^9/L (100,000/µL), transfusion independence
  * CR with incomplete hematologic recovery (CRi): All CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/µL]) or thrombocytopenia (<100 × 10^9/L [100,000/µL])
Time Frame: At the end of Cycle 1 (each cycle is 28 days)
Population: Protocol defined evaluability for participants is defined as completing all Cycle 1 infusions of flotetuzumab (or discontinued treatment due to drug toxicity or disease progression).
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Efficacy as Measured by Number of Participants With CR and CRi
Description: * Complete remission (CR): Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0 × 10^9/L (1000/µL); platelet count ≥100 × 10^9/L (100,000/µL), transfusion independence
  * CR with incomplete hematologic recovery (CRi): All CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/µL]) or thrombocytopenia (<100 × 10^9/L [100,000/µL])
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Population: Protocol defined evaluability for participants is defined as completing all Cycle 1 and 2 infusions of flotetuzumab (or discontinued treatment due to drug toxicity or disease progression) and undergone Cycle 2 Day 28 disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Overall Response Rate
Description: * Defined as partial remission or better
  * PR: All hematologic criteria of CR; decrease of bone marrow blast percentage to 5 to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Population: Protocol defined evaluability for participants is defined as completing all Cycle 1 infusions of flotetuzumab (or discontinued treatment due to drug toxicity or disease progression) and undergone Cycle 2 Day 28 disease assessment (or Cycle 1 Day 28 assessment for patients who only received Cycle 1 of treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 9
Participants | 0

4. Secondary Outcome: Morphologic Leukemia-free State (MLFS) Rate
Description: - MLFS: Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 9
Participants | 0

5. Secondary Outcome: Partial Remission (PR) Rate
Description: - PR: All hematologic criteria of CR; decrease of bone marrow blast percentage to 5 to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 9
Participants | 2

6. Secondary Outcome: Stable Disease (SD) Rate
Description: - SD: Absence of CR(mrd), CR, CRi, PR, MLFS; and criteria for PD not met
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 9
Participants | 3

7. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: * PFS will be calculated as the time from the start of the first dose of study drug until the occurrence of disease progression or death from any cause, respectively
  * Progressive disease: Evidence for an increase in bone marrow blast percentage (>50% over baseline), and/or increase of absolute blast counts in the blood (>50% to >25 × 10^9/L) without differentiation syndrome, or new extramedullary disease
Time Frame: Through completion of follow-up, up to 2 years (median length of 80 days, full range of 11-149 days)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 9
months | 1.14 [0.79 to 2.49]

8. Secondary Outcome: Overall Survival (OS)
Description: -OS will be calculated as the time from the start of the first dose of study drug until the occurrence of death from any cause.
Time Frame: Through completion of follow-up, up to 2 years (median length of 80 days, full range of 11-149 days)
Population: Protocol defined evaluability for participants is defined as having undergone any period of infusion of flotetuzumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
months | 2.66 [1.11 to 4.30]

9. Secondary Outcome: Number of Participants With Adverse Events as Measured by CTCAE v5.0
Time Frame: From start of treatment through 28 days following completion of treatment (median length of 59 days, full range 11-99 days).
Population: Protocol defined evaluability for participants is defined as having undergone any period of infusion of flotetuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
Participants
  Grade 3-5 anemia | 4
  Grade 3-5 febrile neutropenia | 3
  Grade 1-2 sinus tachycardia | 1
  Grade 1-2 adrenal insufficiency | 1
  Grade 1-2 anisocoria | 1
  Grade 1-2 conjunctivitis | 1
  Grade 1-2 scleral hemorrhage | 1
  Grade 1-2 blurred vision | 1
  Grade 1-2 dry eye | 1
  Grade 1-2 melena | 1
  Grade 1-2 white tongue | 1
  Grade 1-2 abdominal distension | 1
  Grade 1-2 abdominal pain | 4
  Grade 3-5 abdominal pain | 1
  Grade 1-2 bloating | 1
  Grade 1-2 constipation | 4
  Grade 1-2 diarrhea | 7
  Grade 1-2 dry mouth | 1
  Grade 1-2 esophageal pain | 1
  Grade 1-2 gastroesophageal reflux disease | 2
  Grade 1-2 hemorrhoids | 1
  Grade 3-5 lower gastrointestinal hemorrhage | 1
  Grade 1-2 mucositis oral | 1
  Grade 1-2 nausea | 5
  Grade 1-2 stomach pain | 1
  Grade 3-5 vomiting | 1
  Grade 1-2 joint pain | 1
  Grade 1-2 chills | 4
  Grade 5 disease progression | 4
  Grade 1-2 edema face | 1
  Grade 3-5 edema face | 1
  Grade 1-2 edema limbs | 3
  Grade 1-2 facial pain | 1
  Grade 1-2 fatigue | 9
  Grade 1-2 fever | 9
  Grade 3-5 fever | 1
  Grade 1-2 generalized edema | 4
  Grade 1-2 injection site reaction | 1
  Grade 1-2 malaise | 3
  Grade 1-2 pain | 4
  Grade 3-5 GvHD of the gut | 1
  Grade 1-2 cytokine release syndrome | 8
  Grade 3-5 cytokine release syndrome | 3
  Grade 1-2 enterococcus | 1
  Grade 1-2staphylococcus aureus | 1
  Grade 1-2 bacteremia | 1
  Grade 1-2 enterocolitis infectious | 1
  Grade 1-2 lung infection | 1
  Grade 3-5 sepsis | 2
  Grade 3-5 sinusitis | 1
  Grade 1-2 viremia | 1
  Grade 1-2 deep tissue injury | 1
  Grade 1-2 fall | 2
  Grade 1-2 infusion related reaction | 1
  Grade 1-2 activated partial thromboplastin time prolonged | 2
  Grade 1-2 alanine aminotransferase increased | 7
  Grade 3-5 alanine aminotransferase increased | 1
  Grade 1-2 alkaline phosphatase increased | 5
  Grade 3-5 alkaline phosphatase increased | 1
  Grade 1-2 aspartate aminotransferase increased | 8
  Grade 1-2 blood bilirubin increased | 8
  Grade 1-2 creatinine increased | 2
  Grade 1-2 INR increased | 6
  Grade 3-5 lymphocyte count decreased | 10
  Grade 3-5 neutrophil count decreased | 7
  Grade 3-5 platelet count decreased | 2
  Grade 1-2 weight gain | 2
  Grade 1-2 white blood cell decreased | 1
  Grade 3-5 white blood cell decreased | 8
  Grade 1-2 anorexia | 1
  Grade 3-5 anorexia | 1
  Grade 1-2 dehydration | 3
  Grade 1-2 hypercalcemia | 1
  Grade 1-2 hyperglycemia | 6
  Grade 3-5 hyperglycemia | 1
  Grade 1-2 hyperkalemia | 1
  Grade 3-5 hyperkalemia | 1
  Grade 1-2 hypermagnesemia | 2
  Grade 1-2 hypernatremia | 3
  Grade 1-2 hyperphosphatemia | 4
  Grade 1-2 hypoalbuminemia | 6
  Grade 3-5 hypoalbuminemia | 3
  Grade 1-2 hypocalcemia | 7
  Grade 3-5 hypocalcemia | 3
  Grade 1-2 hypoglycemia | 1
  Grade 1-2 hypokalemia | 4
  Grade 1-2 hyponatremia | 4
  Grade 1-2 hypophosphatemia | 9
  Grade 1-2 finger stiffness | 1
  Grade 1-2 groin pain | 1
  Grade 1-2 groin swelling | 1
  Grade 1-2 knee pain | 1
  Grade 1-2 shoulder pain | 2
  Grade 1-2 arthralgia | 3
  Grade 3-5 arthralgia | 1
  Grade 1-2 back pain | 2
  Grade 3-5 back pain | 1
  Grade 1-2 bone pain | 2
  Grade 3-5 bone pain | 1
  Grade 1-2 flank pain | 2
  Grade 1-2 generalized muscle weakness | 3
  Grade 1-2 neck pain | 2
  Grade 3-5 neck pain | 1
  Grade 1-2 pain in extremity | 1
  Grade 1-2 expressive aphasia | 1
  Grade 1-2 dizziness | 3
  Grade 3-5 dizziness | 1
  Grade 1-2 dysgeusia | 1
  Grade 1-2 dysphasia | 1
  Grade 1-2 headache | 2
  Grade 1-2 peripheral sensory neuropathy | 1
  Grade 1-2 somnolence | 1
  Grade 3-5 syncope | 1
  Grade 1-2 tremor | 4
  Grade 1-2 incoherent | 1
  Grade 1-2 mental status slightly altered | 1
  Grade 1-2 agitation | 2
  Grade 3-5 agitation | 1
  Grade 1-2 anxiety | 1
  Grade 1-2 confusion | 2
  Grade 3-5 confusion | 1
  Grade 1-2 hallucinations | 2
  Grade 1-2 insomnia | 1
  Grade 1-2 restlessness | 3
  Grade 1-2 acute kidney disease | 1
  Grade 1-2 dieresis | 1
  Grade 1-2 fractional excretion of sodium | 1
  Grade 1-2 dysuria | 1
  Grade 1-2 hematuria | 1
  Grade 1-2 hemoglobinuria | 1
  Grade 1-2 proteinuria | 1
  Grade 1-2 urinary retention | 2
  Grade 1-2 sinus pressure | 1
  Grade 1-2 atelectasis | 1
  Grade 1-2 cough | 2
  Grade 1-2 dyspnea | 5
  Grade 3-5 dyspnea | 2
  Grade 1-2 epistaxis | 2
  Grade 1-2 hypoxia | 4
  Grade 1-2 nasal congestion | 1
  Grade 1-2 productive cough | 2
  Grade 1-2 pulmonary edema | 2
  Grade 3-5 respiratory failure | 2
  Grade 1-2 sinus pain | 1
  Grade 1-2 sore throat | 1
  Grade 1-2 wheezing | 1
  Grade 1-2 oral lesion, left margin of tongue | 1
  Grade 3-5 acute GvHD | 1
  Grade 1-2 pain of skin | 1
  Grade 1-2 pruritus | 2
  Grade 1-2 rash maculo-papular | 2
  Grade 3-5 skin ulceration | 1
  Grade 1-2 flushing | 1
  Grade 1-2 hot flashes | 1
  Grade 1-2 hypotension | 4
  Grade 3-5 hypotension | 1

10. Secondary Outcome: Number of Participants With Cytokine Release Syndrome (CRS) Grading as Measured by ASTCT Consensus Guidelines
Description: * Grade 1:Symptoms are not life threatening and require symptomatic treatment only, e.g., fever, nausea, fatigue, headache, myalgias, malaise
  * Grade 2: Symptoms require and respond to moderate intervention; oxygen requirement < 40% or hypotension responsive to fluids or low-dose of one vasopressor or grade 2 organ toxicity
  * Grade 3: Symptoms require and respond to aggressive intervention; oxygen requirement ≥ 40% or hypotension requiring high-dose vasopressors or multiple vasopressors or grade 3 organ toxicity (except transaminitis) or grade 4 transaminitis
  * Grade 4: Life-threatening symptoms; requirement for ventilator support or grade 4 organ toxicity (excluding transaminitis)
  * Grade 5 Death
Time Frame: Through the end of Cycle 2 (each cycle is 28 days)
Population: Protocol defined evaluability for participants is defined as having undergone any period of infusion of flotetuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
Participants
  Grade 1 | 1
  Grade 2 | 7
  Grade 3 | 3
  Grade 4 | 0
  Grade 5 | 0

11. Secondary Outcome: Number of Participants With Neurotoxicity as Measured by 2019 ASTCT Consensus Guidelines
Time Frame: Through the end of Cycle 2 (each cycle is 28 days)
Population: Protocol defined evaluability for participants is defined as having undergone any period of infusion of flotetuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
Participants | 4

12. Secondary Outcome: Number of Participants With Acute Graft Versus Host Disease (GvHD) as Measured by MAGIC Criteria
Time Frame: Through completion of follow-up, up to 2 years (median length of 80 days, full range of 11-149 days)
Population: Protocol defined evaluability for participants is defined as having undergone any period of infusion of flotetuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
Participants | 1

13. Secondary Outcome: Number of Participants With Chronic Graft Versus Host Disease (GvHD) as Measured by NIH Severity Score
Time Frame: Through completion of follow-up, up to 2 years (median length of 80 days, full range of 11-149 days)
Population: Protocol defined evaluability for participants is defined as having undergone any period of infusion of flotetuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Flotetuzumab
Number analyzed (Participants) | 11
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from start of treatment through 28 days following discontinuation of flotetuzumab (median length of 59 days, full range 11-99 days). All-cause mortality was collected from start of treatment through completion of protocol defined follow-up (median length of 80 days, full range of 11-149 days).
Arm/Group | Flotetuzumab
All-Cause Mortality (participants affected / at risk) | 10/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flotetuzumab (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Disease progression (General disorders) | 4
Cytokine release syndrome (Immune system disorders) | 1
GvHD of the gut (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flotetuzumab (N=11)
Anemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Anisocoria (Eye disorders) | 1
Blurred vision (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Scleral hemorrhage (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Melena (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
White tongue (Gastrointestinal disorders) | 1
Chills (General disorders) | 4
Edema face (General disorders) | 2
Edema limbs (General disorders) | 3
Facial pain (General disorders) | 1
Fatigue (General disorders) | 9
Fever (General disorders) | 10
Generalized edema (General disorders) | 4
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 3
Pain (General disorders) | 4
Cytokine release syndrome (Immune system disorders) | 10
Bacteremia (Infections and infestations) | 1
Enterococcus (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcus aureus (Infections and infestations) | 1
Viremia (Infections and infestations) | 1
Deep tissue injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 8
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 2
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Finger stiffness (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Groin swelling (Musculoskeletal and connective tissue disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Expressive aphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 4
Agitation (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 3
Hallucinations (Psychiatric disorders) | 2
Incoherent (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental status slightly altered (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 3
Acute kidney disease (Renal and urinary disorders) | 1
Dieresis (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Fractional excretion of sodium (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pressure (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acute skin GvHD (rash maculo-papular) (Skin and subcutaneous tissue disorders) | 1
Oral lesion, left margin of tongue (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT04582864/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT04582864/ICF_000.pdf